CLINICAL TRIAL: NCT03768934
Title: A Randomized Controlled Trial of Airtime Incentives to Improve Short Message Service (SMS) Survey Performance in Colombia and Tanzania
Brief Title: Use of Airtime Incentives to Improve Short Message Service Surveys in Colombia and Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: The Bloomberg Family Foundation, Inc. (Other); Ifakara Health Institute (Other); Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318-4.2
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; short message service; incentive
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four airtime amounts: 1) no incentive; 2) 1X incentive; 3) 2X incentive or 4) a lottery incentive, in which one out of every 20 participants will receive the incentive.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No airtime incentive for completing the survey
- 1X Incentive (Experimental): 1X airtime incentive
  Interventions: Other: 1X airtime incentive
- 2X incentive (Experimental): 2X airtime incentive
  Interventions: Other: 2X airtime Incentive
- Lottery Incentive (Experimental): Lottery airtime incentive where odds of winning lottery are 1 out of 20
  Interventions: Other: Lottery airtime incentive

INTERVENTIONS:
Other: 1X airtime incentive — An incentive given in the form of airtime.
  Arms: 1X Incentive
Other: 2X airtime Incentive — An incentive given in the form of airtime.
  Arms: 2X incentive
Other: Lottery airtime incentive — An incentive given in the form of airtime.
  Arms: Lottery Incentive

SUMMARY:
This study evaluates the effect of four different airtime incentive amounts on short message service (SMS) survey cooperation, response, refusal and contact rates, as compared to control group, in Colombia and Tanzania.

DETAILED DESCRIPTION:
Using random digit dialing (RDD) sampling technique, participants were randomized to one of four airtime incentive amounts contingent on them completing the noncommunicable disease risk factor survey. This mobile phone survey will be sent as a short message service (SMS). In SMS surveys, participants use their touch tone key pad to answer written questions. (i.e. If you are male, press 1; If you are female, press 2). This study will be conducted in both Colombia and Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Colombia, conversant in the Spanish language. In Tanzania, conversant in the Swahili language.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2151 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Cooperate Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, cooperation rate is defined as I/(I+P+R) where I is complete interviews, P is partial interviews, and R is refusals and breakoffs.
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, response rate is defined as (I+P)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns.

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, refusal rate is defined as (R)/(I+P+R+eU) where R is refusals and breakoffs, I is complete interviews, P is partial interviews, and eU is the estimated eligible proportion of unknowns.
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, contact rate is defined as (I+P+R)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan A Hyder, PhD, MBBS, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; George W Pariyo, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (2):
- Instituto de Salud Publica Pontificia Universidad Javeriana, Bogotá, D.C., Colombia
- Ifakara Health Institute, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722